CLINICAL TRIAL: NCT03997747
Title: A Study to Assess the Therapeutic Efficacy in Advanced Osteosarcoma Patients In the Clinical Trial of SHR1020-SHR-1210-II-OS (Famitinib and Camrelizumab on Chemo-refractory Osteosarcoma) Based on Genomic Analyses of Tumor Specimens
Brief Title: Cancer Genome Study Using Samples From Patients Treated on Clinical Trial SHR1020-SHR-1210-II-OS
Acronym: CSSG-02
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry); OrigiMed (Industry)
Responsible Party: Sponsor
Other Study IDs: PKUPH-sarcoma 07
Record Dates: First submitted 2019-05-14; First posted 2019-06-25 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Osteosarcoma
Keywords: genomic biomarkers; famitinib; camrelizumab; tumor mutation burden; PD-L1 expression; Tcell-inflamed gene expression profile (GEP)
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tumor samples from patients enrolled on SHR1020-SHR-1210-II-OS before administration of study drug and the first disease progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- comprehensive genomic analysis group: Patients undergo collection of tissue samples for genomic analysis via mass spectrometry, PCR, and microarray. The therapy patients received would not be based on the results of the genomic analysis.
  Interventions: Other: cytology specimen

INTERVENTIONS:
Other: cytology specimen — Biopsy and Genetic: DNA analysis;Genetic: RNA analysis;Genetic: microarray analysis; Genetic: mutation analysis; Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with advanced osteosarcoma refractory to chemotherapy in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to osteosarcma treatment combining anti-angiogenesis tyrosine kinase inhibitors and anti-PD-1 antibody.

PURPOSE: This research study is looking at the cancer genome using tumor samples from patients with advanced stage osteosarcoma treated on clinical trial SHR1020-SHR-1210-II-OS.

DETAILED DESCRIPTION:
OBJECTIVES:

To investigate the clinical relevance of conducting comprehensive molecular analyses on clinically annotated high-quality tumor specimens from patients with advanced stage osteosarcoma.

OUTLINE: This is a single-center study.

Biological specimens are collected from participating clinical site and analyzed by transcription profiling of RNA and microRNA; detection of DNA copy number changes and chromosomal rearrangements; epigenetic modifications analyses; and sequencing of genomic segments, genes, and regulatory regions to assess sequence variation. Clinical information associated with each specimen donor is also collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high-grade osteosarcoma
* refractory to chemotherapy and intended to receive famitinib and camrelizumab following the protocols of SHR1020-SHR-1210-II-OS
* Available tumor tissue samples collected before study drug and after first progression
* Must have matching frozen samples of normal tissue and blood

Exclusion Criteria:

* Patients with concurrent malignancy; patients with prior or concurrent malignancy will be allowed as long as the treating physician considers it unlikely to impact the clinical outcome of the patient
* Serious medical illness including but not limited to uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction or cerebrovascular event with 6 months of registration, history of chronic active hepatitis or history of human immunodeficiency virus (HIV) or an active bacterial infection will not be eligible
* Pregnant or lactating women

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients have histologically proven metastatic or locally advanced osteosarcoma, reviewed by the Pathology Committee of Peking University People's Hospital, and are not amenable to curative-intent surgery. Previous systemic chemotherapy had failed to prevent the exacerbation of disease, including high-dose methotrexate (HD-MTX), doxorubicin (ADM), cisplatin (DDP) with/without ifosfamide (IFO). Tumors have to be measurable with computed tomography scan or magnetic resonance imaging, per RECIST, version 1.1. Patients undergo collection of tissue samples for genomic analysis via mass spectrometry, PCR, and microarray.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
tumor mutation burden | 2 years
  NGS analysis, based on total exon sequencing of the specimen. Identification and characterization of tumor mutation burden.
T cell-inflamed gene expression profile (GEP) | 2 years
  IFN-g-related mRNA profile

SECONDARY OUTCOMES:
single nucleotide variants (SNVs) | 2 years
  NGS analysis, based on total exon sequencing of the specimen
short insertions and deletions (indels) | 2 years
  NGS analysis, based on total exon sequencing of the specimen
copy-number variants (CNVs) | 2 years
  NGS analysis, based on total exon sequencing of the specimen

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D. and Ph.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No